CLINICAL TRIAL: NCT04579653
Title: Effects of Various Non-invasion Stimulation Parameters on Pupil Dilation
Brief Title: Pupillometry and Locus Coeruleus Activation (PuLCA)
Acronym: PuLCA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff who where to run the study left.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201903471
Record Dates: First submitted 2020-08-05; First posted 2020-10-08 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Visual Impairment; Ocular Illness
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: This study has a within-subjects design with a randomization of the order of tVNS administered parameters
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A: Experimental (Experimental): Within-subjects design with a randomization of the order of tVNS administered parameters
  Interventions: Device: transcutaneous electrical nerve stimulation devices
- Group B: Active Comparator (Active Comparator): Within-subjects design with a randomization of the order of tVNS administered parameters
  Interventions: Device: transcutaneous electrical nerve stimulation devices

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation devices — electrical stimulation through surface electrodes
  Other Names: Digitimer DS7A, Ultima Neo, or InTENSity EX4.

SUMMARY:
This project will apply non-invasive, trans-cutaneous vagal nerve stimulation using various stimulation parameters to young, healthy adults to find the optimal set of parameters to elicit pupil response.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speaker with reading and writing proficiency.

Exclusion Criteria:

* Participants with significant visual impairment or ocular illness may be excluded at the discretion of the principal investigator.
* Major medical illnesses including severe neurological illness (e.g. stroke, seizure history), autoimmune disorders, and severe psychiatric diseases (e.g., schizophrenia)
* Any history of brain surgery, tumor, intracranial metal implantation, pacemakers, or other implanted devices.
* Current (i.e. within 48 hours of the session) prescription medication or over-the-counter medication use.
* Illicit alcohol or drug use. Caffeine (e.g, coffee, energy drinks) consumption prior to the visit.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-22 (Estimated); Primary Completion 2023-11-23 (Estimated); Study Completion 2023-11-24 (Estimated)

PRIMARY OUTCOMES:
Ocular response after transcutaneous nerve stimulation | Visit 1 day
  Number of participants with pupil response after transcutaneous nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Porges, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States